CLINICAL TRIAL: NCT01572311
Title: Study of Community Based Dual Task and Aerobic Exercise Intervention on Cognition and Mobility in Older Adults Without Dementia
Brief Title: Dual Task Aerobic Exercise for Older Adults With Cognitive Impairment (HM2)
Acronym: HM2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parkwood Hospital, London, Ontario (Other)
Collaborators: University of Western Ontario, Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Robert Petrella, MD, Principal Investigator, Parkwood Hospital, London, Ontario
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DAE-1234
Record Dates: First submitted 2012-04-03; First posted 2012-04-06 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Cognitive Impairment
Keywords: Aerobic exercise; Cognition; Dual Task; Gait Training; Group-based exercise; Older adults
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Intervention Group (Experimental): For 26 weeks, attend Canadian Centre for Activity and Aging combined classes (75-minute or 60-minute classes, 2 to 3 days/week) and also complete 45 minutes of dual-task gait training (15 minutes for 3 days/week or 22.5 minutes for 2 days/week)
  Interventions: Behavioral: Exercise Intervention
- Exercise Control group (Active Comparator): For 26 weeks, attend Canadian Centre for Activity and Aging combined classes (75-minute or 60-minute classes, 2 to 3 days/week) and also complete 45 minutes of gait training (15 minutes for 3 days/week or 22.5 minutes for 2 days/week). Note: no dual-task challenges during gait training
  Interventions: Behavioral: Exercise Control

INTERVENTIONS:
Behavioral: Exercise Intervention — Goal of 150 minutes of structured exercise/week; minimum of 120 minutes from CCAA classes/week. The 75-minute class includes: 5-minute warm-up; 25 minutes of AE (70-85% maximum heart rate); 5-minute cool-down; 20 minutes of strength training; 5 minutes of core strengthening; 5 minutes of balance training; and 10 minutes of stretching. The 60-minute program is identical except: 15 minutes total for all strength training (including core) and 5 minutes of stretching. Following CCAA classes, participants continue with dual-task gait training where they are required to walk on a special mat with a designated walking pattern (beginner level Square Stepping Exercise) while answering cognitively challenging questions.
  Other Names: Aerobic exercise and dual-task training
  Arms: Exercise Intervention Group
Behavioral: Exercise Control — Goal of 150 minutes of structured exercise/week; minimum of 120 minutes from CCAA classes/week. The 75-minute class includes: 5-minute warm-up; 25 minutes of AE (70-85% maximum heart rate); 5-minute cool-down; 20 minutes of strength training; 5 minutes of core strengthening; 5 minutes of balance training; and 10 minutes of stretching. The 60-minute program is identical except: 15 minutes total for all strength training (including core) and 5 minutes of stretching. Following CCAA classes, participants continue with gait training where they are required to walk on a special mat with a designated walking pattern (beginner level Square Stepping Exercise). This will not include any dual-task challenges.
  Other Names: Aerobic exercise and gait training
  Arms: Exercise Control group

SUMMARY:
The investigators proposed research will establish whether combining aerobic exercise with cognitive challenges is feasible and effective in community dwelling older adults with early signs of cognitive impairment.

DETAILED DESCRIPTION:
To determine the effects of dual-task aerobic exercise training on community dwelling older adults with early signs of cognitive impairment. We will compare an exercise intervention (E-I) versus an exercise control (E-C) group. Each week, both groups will accumulate a minimum of 120 minutes of exercise (target 150 minutes) from community-based group classes (50 minutes of aerobic exercise) and also complete 45 minutes of beginner-level Square Stepping Exercise (SSE). The E-I group will also answer cognitively challenging questions while doing SSE (dual-task training). This study will determine whether a combined multiple modality (primary component being aerobic exercise) and dual-task exercise program is both feasible and effective for improving cognitive and mobility status, as well as vascular compliance, in older adults who may be at risk for cognitive and mobility decline.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female 55-90 years old.
* Montreal Cognitive Assessment score ≤27
* Preserved Instrumental Activities of Daily Living (based on Lawton-Brody Instrumental Activities of Daily Living Sale)

Exclusion Criteria:

* Dementia (i.e., Mini-Mental Examination score <24 or self-reported physician diagnosis)
* Major Depression (>=16 on the Center for Epidemiologic Studies - Depression Scale combined with clinical judgment by primary study physician)
* Other neurological or psychiatric disorders
* Recent history of severe cardiovascular conditions
* Significant orthopedic conditions
* Have blood pressure >180/100 mmHg or <100/60 mmHg
* Unable to comprehend questionnaire material/study procedures

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-06; Primary Completion 2013-11 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Global cognitive functioning | 26 weeks
  Four standardized domain-specific composite scores were averaged to create this standardized global cognitive functioning score (incorporates executive function, processing speed, verbal learning and memory, and verbal fluency.

SECONDARY OUTCOMES:
Global cognitive functioning | 12 & 52 weeks
  Four standardized domain-specific composite scores were averaged to create this standardized global cognitive functioning score (incorporates executive function, processing speed, verbal learning and memory, and verbal fluency.
Executive Function/Mental Flexibility | 12, 26, and 52 weeks
  Standardized scores from seconds to complete Trail Making Test Part A and Trail Making Test Part B averaged to create this standardized composite score
Processing Speed | 12, 26 and 52 weeks
  Standardized score from the Digit-Symbol Substitution Test (total correct responses)
Verbal Learning and Memory | 12, 26 and 52 weeks
  Standardized scores from Auditory Verbal Learning Test (number of words learned and number of words recalled) were averaged to create this standardized composite score
Verbal Fluency | 12, 26 and 52 weeks
  Standardized scores from semantic (number of animals) and phonemic (number of words starting with C) were averaged to create this standardized composite score
Gait variability (step length) under dual-task conditions | 12, 26 and 52 weeks
  Gait variability is the stride-to-stride fluctuations of the way someone walks and will be calculated as coefficient of variation of step length (SD/mean x 100). Measured with GAITRite system.
Gait variability (step length) under single-task conditions | 12, 26 and 52 weeks
  Gait variability is the stride-to-stride fluctuations of the way someone walks and will be calculated as coefficient of variation of step length (SD/mean x 100). Measured with GAITRite system.
Gait speed under dual-task conditions | 12, 26 and 52 weeks
  Average walking speed measured with GAITRite system
Gait speed under single-task conditions | 12, 26 and 52 weeks
  Average walking speed measured with GAITRite system
Double support (seconds and % gait cycle time) under dual-task conditions | 12, 26 and 52 weeks
  Initial double support occurs from heel contact of one footfall to toe-off of the opposite footfall. Terminal double support occurs from opposite footfall heel strike to support footfall toe-off.Total double support is the sum of the initial double support added to the terminal double support. It is measured in seconds (sec) and also expressed as a percent of the Gait Cycle time for the same foot. Measured with GAITRite system
Double support (seconds and % gait cycle time) under single-task conditions | 12, 26 and 52 weeks
  Initial double support occurs from heel contact of one footfall to toe-off of the opposite footfall. Terminal double support occurs from opposite footfall heel strike to support footfall toe-off.Total double support is the sum of the initial double support added to the terminal double support. It is measured in seconds (sec) and also expressed as a percent of the Gait Cycle time for the same foot. Measured with GAITRite system
Step length under dual-task conditions | 12, 26 and 52 weeks
  Mean step length measured with GAITRite system
Step length under single-task conditions | 12, 26 and 52 weeks
  Mean step length measured with GAITRite system
Carotid artery compliance | 12, 26 and 52 weeks
  Measured from non-invasive vascular assessment with B-mode Ultrasound over the carotid artery (in the neck)
Carotid artery Intima-media thickness (IMT) | 12, 26 and 52 weeks
  Measured from non-invasive vascular assessment with B-mode Ultrasound over the carotid artery (in the neck)
Ambulatory systolic blood pressure | 12, 26 and 52 weeks
  Average systolic blood pressure over a 24-hour time frame
Clinic systolic blood pressure | 12, 26 and 52 weeks
  Average systolic blood pressure from final 2 (out of 3) readings
Ambulatory diastolic blood pressure | 12, 26 and 52 weeks
  Average diastolic blood pressure over a 24-hour time frame
Clinic diastolic blood pressure | 12, 26 and 52 weeks
  Average diastolic blood pressure from final 2 (out of 3) readings
Total balance score | 12, 26, and 52 weeks
  Total balance score calculated from the Fullerton Advanced Balance Scale
Total Falls Self-Efficacy score | 12, 26, and 52 weeks
  Total falls self-efficiacy score calculated from the Falls Self-Efficacy International (FES-I) scale

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Petrella, MD., PhD., Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Aging, Rehabilitation and Geriatric Care Research Center, London, Ontario, Canada

REFERENCES:
- [Derived] Gill DP, Gregory MA, Zou G, Liu-Ambrose T, Shigematsu R, Hachinski V, Fitzgerald C, Petrella RJ. The Healthy Mind, Healthy Mobility Trial: A Novel Exercise Program for Older Adults. Med Sci Sports Exerc. 2016 Feb;48(2):297-306. doi: 10.1249/MSS.0000000000000758. PMID 26285025